CLINICAL TRIAL: NCT04475211
Title: Predictors of Mortality at Day 28 of Patients Treated at Lille University Hospital for COVID-19
Brief Title: LILLE COVID RESEARCH NETWORK (Covid-19)
Acronym: LICORNE
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_54; 2020-A01514-35 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-07-10; First posted 2020-07-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Sars-CoV2
Keywords: COVID-19; fatality rate; Inflammatory and autoimmune processes; severity; clinical features; diagnostic (qRT-PCR or serology) methods; thrombosis; co-infection
MeSH Terms: conditions — COVID-19; Disease; Thrombosis; Coinfection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood, plasma, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Lille University Hospital developped a research objective common to all the services which took care of patients, "suspected patient", "possible case", "probable case" or "confirmed case" infected with SARS-CoV-2 by constituting a prospective and a retrospective observational cohort which allowed pooling and sharing the resources and data collected. In the next two years the prospective cohort will allow to continue inclusions in a standardized way mainly for the constitution of a negative control group (excluded cases), to collect biological samples which had not been collected in the retrospective cohort so that the pathophysiology of the COVID-19 will be better apprehended as for example the inflammatory response to the viral infection. Finally in case of a second epidemic wave in the Hauts De France, it seems essential to have a defined research protocol which had already received all the necessary authorizations to guarantee cutting-edge (or quality ) research in a center like the Lille University Hospital.The aim objective of this study is to identify predictive factors of mortality to day 28 infection to SARS-CoV-2 for patients under medical care for the COVID-19 in the Lille University Hospital thanks to the constitution of an epidemiological, clinical, biological, immunological, genetic, microbiological, anatomopathologic, radiological, therapeutic database and so record the results of functional exploration exams.

DETAILED DESCRIPTION:
This is a retrospective and prospective observational monocentric cohort study designed to identify predictors of mortality on day 28 in patients treated at the Lille University Hospital for COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* All adult "suspect patient", "possible case", "probable case" or "confirmed case" of an SARS-CoV-2 infection admitted to Lille University Hospital.

Exclusion Criteria:

* Minor patient Patient under guardianship or curatorship Refusal to participate in the study Patient for whom the collection of genetic non-opposition or consent is impossible because of a language barrier with the patient himself or herself or with his or her trusted person or close family.

Patient for whom the collection of genetic non-opposition or consent is impossible because of his or her state of health at the time of inclusion in the study and for whom the trusted person or close family member opposes participation in the study.

Translated with www.DeepL.com/Translator (free version)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult "suspect patient", "possible case", "probable case" or "confirmed case" of an SARS-CoV-2 infection admitted to Lille University Hospital.
Sampling Method: Probability Sample
Enrollment: 757 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Number of patients "confirmed cases" of SARS-CoV-2 infection who died at D28 of inclusion | At 28 days
  Identify predictors of mortality at day 28 in patients treated at the Lille University Hospital for COVID-19

SECONDARY OUTCOMES:
Correlation between Infection characteristics of patients at inclusion and all predictors for Covid-19 | At inclusion (day 0)
  Describe, at inclusion, the epidemiological, clinical, biological, immunological, genetic, microbiological, radiological, therapeutic characteristics and the results of functional explorations of patients hospitalized in our center with SARS-CoV-2 infection.
Correlation between evolution infection characteristics of patients during stay of hospitalisation and all predictors for Covid-19 | At inclusion ( day 0) ,at day 1 , day3±1, Day 5±1, day 7±1, day 9±2, day14±2, day30±3, at months 3±7 days and at months6±7days or until death
  Describe the evolution of the characteristics the epidemiological, clinical, biological, immunological, genetic, microbiological, anatomopathological, radiological, therapeutic characteristics and the results of functional explorations of patients hospitalized in our center with SARS-CoV-2 infection.
Positivity for Covid-19 patients performed and all predictors for Covid-19 | At inclusion (day 0)
  The diagnosis of disease is excluded or confirmed by qRT-PCR SARS-CoV-2 (respiratory samples, blood, stool...) and/or serology.
Correlation between hospitalisation and all predictors for Covid-19 | At inclusion( Day 0)
  Identify epidemiological, clinical, radiological, biological, immunological and genetic predictors of hospitalization in patients with SARS-CoV-2 infection.
Correlation between risk factors measured at D0 for severe CoV-2 SARS infection and all predictors for Covid-19 | At 28 day
  Identify epidemiological, clinical, radiological, biological, immunological and genetic predictors of sévère SARS-CoV-2 infection.
Correlation between overall survival at Day 28 and all predictors for Covid-19 | At 28 day
  Identify epidemiological, clinical, radiological, biological, immunological, genetic and therapeutic predictors of survival in patients with SARS-CoV-2 infection.
Cumulative incidence of at least one complication related to COVID 19 | during hospitalization or during outpatient follow-up of "confirmed case" patients at Lille University Hospital (maximum observation period 6 months).
  Death is a concurrent risk.
Cumulative incidence of the thrombosis complication related to COVID 19 | during hospitalization or during outpatient follow-up of "confirmed case" patients at Lille University Hospital (maximum observation period 6 months).
  Death is a concurrent risk.
All type of co-infections | At 6 months
  Describe viral (other than SARS-CoV-2), bacterial and fungal co-infections in patients admitted for COVID disease 19. The appropriateness of the co-infection search is at the discretion of the clinician to fit the patient's history and clinical presentation
Alteration of microbiota | At 6 months
  alterations in respiratory and digestive microbiotes and their evolution potentially associated with bacterial or fungal superinfection in the most severe patients
Biobanking for further analyses such as SARS-CoV2 studies | At 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Charlotte CHOPIN, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chr Lille, Lille, France

IPD SHARING:
Plan to Share IPD: Undecided